CLINICAL TRIAL: NCT02694822
Title: A Phase 1/2, Open-Label, Multicenter Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of an Anti-CTLA-4 Human Monoclonal Antibody (AGEN1884) in Subjects With Advanced or Refractory Cancer and in Subjects Who Have Progressed During Treatment With a PD-1/PD-L1 Inhibitor as Their Most Recent Therapy
Brief Title: AGEN1884, an Anti-CTLA-4 Human Monoclonal Antibody in Participants With Advanced or Refractory Cancer and Who Have Progressed With PD-1/PD-L1 Inhibitor as Their Most Recent Therapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-500-01
Record Dates: First submitted 2016-02-12; First posted 2016-03-01 (Estimated); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Advanced Solid Cancers; Advanced Solid Cancers Refractory to PD-1 and PD-L1 Therapies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zalifrelimab (Experimental): Participants received zalifrelimab intravenously.
  Interventions: Drug: Zalifrelimab

INTERVENTIONS:
Drug: Zalifrelimab — An anti-CTLA-4 monoclonal antibody.
  Other Names: AGEN1884

SUMMARY:
This is an open-label, Phase 1/2, multicenter study to evaluate the safety, pharmacokinetics, and pharmacodynamics of an anti-cytotoxic T lymphocyte-associated protein-4 (CTLA-4) human monoclonal antibody (zalifrelimab) in participants with advanced or refractory cancer and in participants who have progressed during treatment with a programmed cell death protein-1/programmed cell death ligand-1 (PD-1/PD-L1) inhibitor as their most recent therapy.

The phase 1 portion of the study has been completed; it enrolled adult participants with refractory, advanced cancer in a 3+3 dose escalation cohort.

The phase 2 portion consisted of 51 participants who progressed during treatment with an approved or investigational PD-1/PD-L1 inhibitor as their most recent therapy (2-6 weeks prior to first dose of study drug).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. ≥18 years of age.
3. Histological or cytological diagnosis of solid cancer or lymphoma that is considered incurable and without therapies with established benefit. Biopsy is not necessary for participants with known prior diagnosis, and clinical or radiographic evidence of recurrence. For Phase 2 only: Participants who experienced documented disease progression during treatment with an approved or investigational PD-1/PD-L1 inhibitor as their most recent therapy (2-6 weeks prior to first dose of study drug). This cohort includes participants with histological diagnoses of hepatocellular carcinoma (HCC) (not including atypical histology such as cholangiocarcinoma mix or fibrolamellar hepatocellular carcinoma) who experienced documented disease progression during treatment with an approved or investigational PD-1/PD-L1 inhibitor as their most recent therapy (2-6 weeks prior to first dose of study drug).
4. Eastern Cooperative Oncology Group (ECOG) score of 0 or 1.
5. Participants in Phase 2 with HCC should have a Child-Pugh score of A or B7 with no encephalopathy or ascites.
6. Life expectancy ≥12 weeks.
7. Adequate cardiac function (New York Heart Association [NYHA] class ≤II).
8. Adequate organ function, defined as absolute neutrophil count (ANC) ≥1,500×10^6/liter (L), absolute lymphocyte count ≥500/cubic millimeters (mm^3), hemoglobin ≥8.0 grams/deciliter (g/dL), and platelet count ≥100,000×10^6/mm^3 without blood growth factors or without transfusions within 1 week of first dose. For participants in Phase 2 with HCC: Platelet count ≥60×10^6/mm^3 and ANC ≥1,000×10^6/L are acceptable provided that the principal investigator assesses these abnormalities as due to liver disease.
9. Adequate liver function, defined as aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5× institutional upper limit of normal (ULN), and bilirubin ≤1.5 milligrams/deciliter (mg/dL) × ULN. For participants in Phase 2 with HCC: AST and ALT ≤5 × ULN, bilirubin ≤2 mg/dL × ULN, and albumin ≥2.8 mg/dL.
10. Adequate renal function, defined as estimated creatinine clearance ≥50 milliliters/minute according to Cockcroft-Gault formula, or measured 24-hour creatinine clearance (or local institutional standard method).
11. Adequate coagulation defined by international normalized ratio (INR) or prothrombin time (PT) ≤1.5× ULN (unless the participant is receiving anticoagulant therapy); and activated partial thromboplastin time ≤1.5× ULN (unless the participant is receiving anticoagulant therapy). Participants in Phase 2 with HCC can have an INR ≤2.3× ULN. Note: Participants in Phase 2 with HCC and on anticoagulant treatment would have an assigned value of 1 point when scoring PT/INR so the overall Child-Pugh score is not adversely affected.
12. Female participants of childbearing potential and fertile male participants must agree to use adequate contraception or abstain from sexual activity from the time of consent through 90 days after the end of study drug. Adequate contraception includes condoms with contraceptive foam; oral, implantable, or injectable contraceptives; contraceptive patch; intrauterine device; diaphragm with spermicidal gel; or a sexual partner who is surgically sterilized or postmenopausal. Note: Abstinence is acceptable if this is the established and preferred contraception for the participant.
13. In the expansion phase, all participants must provide a sufficient and adequate formalin-fixed paraffin embedded (FFPE) tumor tissue sample preferably collected after progression on the last therapy and/or collected at screening, if clinically feasible. If a recent biopsy is not available, an archival FFPE sample should be provided from a site not previously irradiated. If no tumor tissue is available, a fresh biopsy will be required if clinically feasible.

Exclusion Criteria

1. Other malignancies treated within the last 5 years, except in situ cervix carcinoma or non-melanoma skin cancer.
2. Other form(s) of antineoplastic therapy anticipated during the period of the study.
3. Previous severe hypersensitivity reaction to another fully human monoclonal antibody or severe reaction to immuno-oncology agents, such as colitis or pneumonitis requiring treatment with steroids.
4. History of interstitial lung disease.
5. Primary or secondary immunodeficiency, including immunosuppressive disease, autoimmune disease (including autoimmune endocrinopathies), or usage of immunosuppressive medications.

   Note: Participants with diabetes type 1, vitiligo, psoriasis, hypo-, or hyperthyroid disease not requiring immunosuppressive treatment are eligible. Participants with Type 2 diabetes mellitus are allowed.
6. Participants with a known history of human immunodeficiency virus 1 and 2, human T lymphotropic virus 1.

   Participants in Phase 2 with HCC: Participants with active hepatitis B infection who are receiving effective antiviral therapy are permitted. Participants with active hepatitis C infection are allowed (antiviral therapy not required).
7. Administration of anticancer medications or investigational drugs within the following intervals before the first administration of study drug: a. ≤14 days for chemotherapy, targeted small molecule therapy, or radiation therapy. Participants must also not have had radiation pneumonitis as a result of treatment and cannot participate in the study if they are on chronic corticosteroids for radiation pneumonitis. A 1-week washout is permitted for palliative radiation to non-central nervous system (CNS) disease, with medical monitor approval.

   Note: Bisphosphonates and denosumab are permitted medications. b. ≤14 days for prior immunotherapy. Participants in the dose escalation cohorts are excluded if they have received prior checkpoint inhibitors, costimulatory agonists, or immune modulating therapy except as described below. Once a dose level is determined to be safe by the safety review committee, participants will be allowed to enroll in dose-level expansion cohorts if they have received other non-CTLA-4 targeting immunotherapies.

   c. Participants enrolling in Phase 2 must have cancer that has progressed after prior treatment with an approved or investigational PD-1/PD-L1 inhibitor as their most recent therapy (2-6 weeks prior to first dose of study drug). The minimum requirement of 2 weeks (14 days) from prior anti-PD-1/PD-L1 therapy is to allow resolution of any lower-grade (≤2) adverse events observed with the therapy. If the investigator feels the participant has tolerated prior anti-PD-1/PD-L1 therapy well, then treatment with study agent may begin sooner.

   d. ≤7 days for prior corticosteroid treatment, with the following exceptions:
   * Use of an inhaled or topical corticosteroid is permitted.
   * Corticosteroid premedication for radiographic imaging for dye allergies is permitted.
   * Use of physiologic corticosteroid replacement therapy may be approved after consultation with the medical monitor. e. ≤21 days for prior monoclonal antibody used for anticancer therapy, with the exception of denosumab. This does not apply to participants being enrolled in Phase 2, who have received a PD-1/PD-L1 inhibitor as their most recent therapy (2-6 weeks prior to first dose of study drug; see above).

     f. ≤7 days for immunosuppressive-based treatment for any reason, with the exceptions noted above for prior corticosteroid treatment (exclusion criterion d).

     g. ≤21 days or 5 half-lives before first dose of study treatment for all other investigational study drugs or devices. For investigational agents with long half- lives (for example, >5 days), enrollment before the fifth half-life requires medical monitor approval.

     h. For participants in Phase 2 with HCC <6 weeks for prior locoregional therapy to the liver, for example, transcatheter chemoembolization, radiation, surgery, or radioembolization.
8. Has not recovered to grade ≤1 from toxic effects of prior therapy and/or complications from prior surgical intervention before starting therapy.

   Note: Participants with grade ≤2 neuropathy and alopecia are an exception and may enroll.
9. Uncontrolled infection or other serious medical illnesses.
10. History or presence of an abnormal electrocardiogram that, in the investigator's opinion, is clinically meaningful.
11. Any medical conditions that, in the opinion of the investigator, would preclude use of AGEN1884, including AGEN1884 hypersensitivity.
12. Women who are pregnant or breastfeeding.
13. Concurrent participation in other investigational drug trials.
14. Has a CNS tumor, metastasis(es), and/or carcinomatous meningitis identified either on the baseline brain imaging obtained during the screening period or identified prior to consent. Note: Participants with history of brain metastases that have been treated may participate provided they show evidence of stable supra-tentorial lesions are obtained after treatment to the brain metastases. These imaging scans should both be obtained ≥4 weeks apart). In addition, any neurologic symptoms that developed either as a result of the brain metastases or their treatment must have returned to baseline or resolved. For individuals who received steroids as part of brain metastases treatment, steroids must be discontinued ≥7 days prior to first dose of study drug.
15. For participants in Phase 2 with HCC, the following exclusions also apply:

    1. Recent encephalopathy episodes in the last 6 months.
    2. Recent (within the last 6 months) gastro-esophageal varices bleeding.
    3. Participant whose tumors have cardiac involvement, as determined by imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Agenus Inc.
Locations (11):
- United States (11):
  - City of Hope National Medical Center, Duarte, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - University of Miami Miller School of Medicine, Miami, Florida
  - Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - Ochsner Cancer Institute, New Orleans, Louisiana
  - Atlantic Health System/Morristown Medical Center, Morristown, New Jersey
  - Levine Cancer Institute, Charlotte, North Carolina
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Texas Oncology - Austin Midtown, Austin, Texas
  - Texas Oncology, Tyler Texas, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: Zalifrelimab Dose 1: Participants received zalifrelimab (0.1 milligrams/kilogram [mg/kg]) intravenously (IV) every 3 weeks (Q3W).
- Phase 1: Zalifrelimab Dose 2: Participants received zalifrelimab (0.3 mg/kg) IV Q3W.
- Phase 1: Zalifrelimab Dose 3; Phase 2: Zalifrelimab: Participants received zalifrelimab (1.0 mg/kg) IV Q3W.
- Phase 1: Zalifrelimab Dose 4: Participants received zalifrelimab (3.0 mg/kg) IV Q3W.
- Phase 1: Zalifrelimab Dose 5: Participants received zalifrelimab (6.0 mg/kg) IV Q3W.
Period: Phase 1
Arm/Group | Phase 1: Zalifrelimab Dose 1 | Phase 1: Zalifrelimab Dose 2 | Phase 1: Zalifrelimab Dose 3 | Phase 1: Zalifrelimab Dose 4 | Phase 1: Zalifrelimab Dose 5 | Phase 2: Zalifrelimab
Started | 5 | 3 | 10 | 15 | 5 | 0
Received at Least 1 Dose of Study Drug (Safety Analysis Set) | 5 | 3 | 10 | 15 | 5 | 0
Completed | 1 | 0 | 0 | 1 | 1 | 0
Not Completed | 4 | 3 | 10 | 14 | 4 | 0
Not completed — Death | 2 | 1 | 6 | 6 | 3 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 4 | 8 | 1 | 0
Period: Phase 2
Arm/Group | Phase 1: Zalifrelimab Dose 1 | Phase 1: Zalifrelimab Dose 2 | Phase 1: Zalifrelimab Dose 3 | Phase 1: Zalifrelimab Dose 4 | Phase 1: Zalifrelimab Dose 5 | Phase 2: Zalifrelimab
Started | 0 (Phase 1 participants did not continue into Phase 2.) | 0 | 0 | 0 (Phase 1 participants did not continue into Phase 2.) | 0 (Phase 1 participants did not continue into Phase 2.) | 51 (Phase 2 participants enrolled separately from Phase 1.)
Received at Least 1 Dose of Study Drug (Safety Analysis Set) | 0 | 0 | 0 | 0 | 0 | 51
Completed | 0 | 0 | 0 | 0 | 0 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 43
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 26
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 13
Not completed — Administrative Study Closure | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Participant Transferred to Another Site | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all participants who received at least 1 dose of zalifrelimab.
Groups:
- Phase 1: Zalifrelimab Dose 1: Participants received zalifrelimab (0.1 mg/kg) IV Q3W.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Zalifrelimab Dose 1 | Phase 1: Zalifrelimab Dose 2 | Phase 1: Zalifrelimab Dose 3 | Phase 1: Zalifrelimab Dose 4 | Phase 1: Zalifrelimab Dose 5 | Phase 2: Zalifrelimab | Total
Number analyzed (Participants) | 5 | 3 | 10 | 15 | 5 | 51 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 6 | 7 | 5 | 30 | 55
  >=65 years | 0 | 1 | 4 | 8 | 0 | 21 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 7 | 8 | 3 | 19 | 41
  Male | 3 | 1 | 3 | 7 | 2 | 32 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 3 | 4 | 0 | 5 | 14
  Not Hispanic or Latino | 4 | 2 | 7 | 11 | 5 | 44 | 73
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 3 | 0 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 2 | 0 | 5 | 8
  White | 4 | 3 | 9 | 9 | 5 | 39 | 69
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Dose-limiting Toxicities (DLTs) of Zalifrelimab
Description: A DLT was defined as a Grade ≥3 adverse drug reaction (ADR), according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5, occurring in the DLT evaluation period (28 days after the initial administration of zalifrelimab). An ADR was defined as all noxious and unintended responses to a medicinal product, related to any dose.
Time Frame: Up to 28 days
Population: DLT Evaluable Analysis Set: all participants within the dose escalation (Phase 1) cohorts who received ≥2 doses of zalifrelimab at their assigned dose level and completed the DLT evaluation period of 28 days, or all participants within the dose escalation cohort who received ≥1 dose of zalifrelimab and experienced a DLT. As pre-specified, data were collected and are reported for Phase 1 only.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Zalifrelimab Dose 1 | Phase 1: Zalifrelimab Dose 2 | Phase 1: Zalifrelimab Dose 3 | Phase 1: Zalifrelimab Dose 4 | Phase 1: Zalifrelimab Dose 5
Number analyzed (Participants) | 5 | 3 | 10 | 15 | 5
Participants | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Phase 1 and Phase 2: Number of Participants Experiencing Any Treatment-related Adverse Events
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that did not necessarily have a causal relationship with this treatment. A treatment-related AE was one in which a causal relationship between the medicinal product and the AE was at least a reasonable possibility and could not be ruled out. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to 6 years
Population: Safety Analysis Set: all participants who received at least 1 dose of zalifrelimab.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Zalifrelimab Dose 1 | Phase 1: Zalifrelimab Dose 2 | Phase 1: Zalifrelimab Dose 3 | Phase 1: Zalifrelimab Dose 4 | Phase 1: Zalifrelimab Dose 5 | Phase 2: Zalifrelimab
Number analyzed (Participants) | 5 | 3 | 10 | 15 | 5 | 51
Participants | 3 | 2 | 6 | 12 | 4 | 31

3. Primary Outcome: Phase 1: Maximum Drug Concentration (Cmax) of Zalifrelimab
Description: Blood samples were collected at designated timepoints to characterize Cmax of serum zalifrelimab following IV infusion in participants with metastatic or locally advanced solid tumors. Data reported as micrograms/milliliter (ug/mL).
Time Frame: Day 1 of Cycle 1 (21 days/cycle)
Population: Pharmacokinetics Analysis Set: all participants who received at least 1 dose of zalifrelimab. As pre-specified, data were collected and are reported for Phase 1 only.
Measure: Median (Standard Error); unit: ug/mL
Arm/Group | Phase 1: Zalifrelimab Dose 1 | Phase 1: Zalifrelimab Dose 2 | Phase 1: Zalifrelimab Dose 3 | Phase 1: Zalifrelimab Dose 4 | Phase 1: Zalifrelimab Dose 5
Number analyzed (Participants) | 5 | 3 | 10 | 15 | 5
ug/mL | 1.95 (0.30946) | 7.15 (1.3635) | 23.1 (1.2891) | 63.5 (9.4314) | 120 (18.075)

4. Primary Outcome: Phase 1: Area Under the Drug Concentration-time Curve From 0 to 21 Days (AUC0-21d) of Zalifrelimab
Description: Blood samples were collected at designated timepoints to characterize AUC0-21d of serum zalifrelimab following IV infusion in participants with metastatic or locally advanced solid tumors. Data reported as hour times ug/mL (hour*ug/mL).
Time Frame: Day 1 of Cycle 1 (21 days/cycle)
Population: as for outcome 3
Measure: Median (Standard Error); unit: hour*ug/mL
Arm/Group | Phase 1: Zalifrelimab Dose 1 | Phase 1: Zalifrelimab Dose 2 | Phase 1: Zalifrelimab Dose 3 | Phase 1: Zalifrelimab Dose 4 | Phase 1: Zalifrelimab Dose 5
Number analyzed (Participants) | 5 | 3 | 10 | 15 | 5
hour*ug/mL | 317 (51.897) | 1522 (246.42) | 3915 (964.89) | 11390 (964.89) | 18803 (2370.77)

5. Secondary Outcome: Phase 1 and Phase 2: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR) as determined by radiographic disease assessments per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1). BOR was defined as the best response recorded from the start of treatment until disease progression/recurrence; any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeters. CR was defined as disappearance of all target lesions, and PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 6 years
Population: Safety Analysis Set: all participants who received at least 1 dose of zalifrelimab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: Zalifrelimab Dose 1 | Phase 1: Zalifrelimab Dose 2 | Phase 1: Zalifrelimab Dose 3 | Phase 1: Zalifrelimab Dose 4 | Phase 1: Zalifrelimab Dose 5 | Phase 2: Zalifrelimab
Number analyzed (Participants) | 5 | 3 | 10 | 15 | 5 | 51
percentage of participants | 20.0 [0.5 to 71.6] | 0 [0.0 to 70.8] | 0 [0.0 to 30.9] | 0 [0.0 to 21.8] | 0 [0.0 to 52.2] | 5.9 [2.0 to 15.9]

6. Secondary Outcome: Phase 1 and Phase 2: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants who had a confirmed response (CR or PR) or stable disease (SD) without progressive disease (PD). SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that is the smallest on study).
Time Frame: Up to 6 years
Population: Safety Analysis Set: all participants who received at least 1 dose of zalifrelimab. Here, 'Overall Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: Zalifrelimab Dose 1 | Phase 1: Zalifrelimab Dose 2 | Phase 1: Zalifrelimab Dose 3 | Phase 1: Zalifrelimab Dose 4 | Phase 1: Zalifrelimab Dose 5 | Phase 2: Zalifrelimab
Number analyzed (Participants) | 5 | 3 | 10 | 15 | 5 | 51
percentage of participants | 20.0 [0.5 to 71.6] | 33.3 [0.8 to 90.6] | 0 [0.0 to 30.9] | 6.7 [0.2 to 32.0] | 0 [0.0 to 52.2] | 37.3 [25.3 to 51.0]

7. Secondary Outcome: Phase 1 and Phase 2: Duration of Response (DOR)
Description: DOR was defined as the interval from which the date measurement criteria were met for CR or PR (whichever was first recorded) until the earliest date of disease progression, as determined by investigator assessment of objective radiographic disease assessments per RECIST v1.1, or death due to any cause, if occurring sooner than progression.
Time Frame: Up to 6 years
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 1: Zalifrelimab Dose 1 | Phase 1: Zalifrelimab Dose 2 | Phase 1: Zalifrelimab Dose 3 | Phase 1: Zalifrelimab Dose 4 | Phase 1: Zalifrelimab Dose 5 | Phase 2: Zalifrelimab
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 3
weeks | NA [NA to NA] — DOR not reached during Phase 1 due to an insufficient number of participants with events. |  |  |  |  | NA [NA to NA] — DOR not reached during Phase 2 due to an insufficient number of participants with events.

8. Secondary Outcome: Phase 1: Progression-free Survival (PFS)
Description: PFS was defined as the interval from the date of first dose of investigational agent until the earliest date of PD, as determined by independent endpoint review committee assessment of objective radiographic disease assessments per RECIST v1.1, or death due to any cause if occurring sooner than progression.
Time Frame: Up to 6 years
Population: Safety Analysis Set: all participants who received at least 1 dose of zalifrelimab. Here, 'Overall Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure in Phase 1.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 1: Zalifrelimab Dose 1 | Phase 1: Zalifrelimab Dose 2 | Phase 1: Zalifrelimab Dose 3 | Phase 1: Zalifrelimab Dose 4 | Phase 1: Zalifrelimab Dose 5
Number analyzed (Participants) | 5 | 3 | 10 | 15 | 5
weeks | NA [3.143 to NA] — Values were non-estimable (insufficient number of participants with events). A lower confidence interval value is reported only since the survival curve crossed 0.5 probability. Only 1 participant experienced the event. The other participants were censored. | 11.000 [4.429 to NA] — Values were non-estimable (insufficient number of participants with events). | 10.429 [5.286 to 12.429] | 11.143 [7.143 to 16.286] | 5.714 [2.571 to NA] — Values were non-estimable (insufficient number of participants with events).

9. Secondary Outcome: Phase 2: PFS
Description: as for outcome 8
Time Frame: Up to 6 years
Population: Safety Analysis Set: all participants who received at least 1 dose of zalifrelimab.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Zalifrelimab
Number analyzed (Participants) | 51
months | 2.0 [1.4 to 2.9]

10. Secondary Outcome: Phase 1: Overall Survival (OS)
Description: OS was defined as the interval from the date of first dose of investigational agent until the date of death. For participants who did not die, OS was censored at last contact date.
Time Frame: Up to 6 years
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 1: Zalifrelimab Dose 1 | Phase 1: Zalifrelimab Dose 2 | Phase 1: Zalifrelimab Dose 3 | Phase 1: Zalifrelimab Dose 4 | Phase 1: Zalifrelimab Dose 5
Number analyzed (Participants) | 5 | 3 | 10 | 15 | 5
weeks | NA [17.429 to NA] — Values were non-estimable (insufficient number of participants with events). A lower confidence interval value is reported only since the survival curve crossed 0.5 probability. Only 2 participants experienced the event. The other participants were censored. | 71.143 [NA to NA] — Values were non-estimable (insufficient number of participants with events). A median value is reported only since the survival curve crossed 0.5 probability. Only 1 participant experienced the event. The other participants were censored. | 20.429 [2.000 to 49.857] | 70.571 [9.857 to NA] — Values were non-estimable (insufficient number of participants with events). | 15.000 [4.857 to NA] — Values were non-estimable (insufficient number of participants with events).

11. Secondary Outcome: Phase 2: OS
Description: as for outcome 10
Time Frame: Up to 6 years
Population: Safety Analysis Set: all participants who received at least 1 dose of zalifrelimab.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Zalifrelimab
Number analyzed (Participants) | 51
months | 16.8 [5.7 to 25.6]

ADVERSE EVENTS:
Time Frame: From Day 1 to the end of study (6 years)
Description: All reported safety data based upon the Safety Analysis Set: all participants who received at least 1 dose of zalifrelimab.
Arm/Group | Phase 1: Zalifrelimab Dose 1 | Phase 1: Zalifrelimab Dose 2 | Phase 1: Zalifrelimab Dose 3 | Phase 1: Zalifrelimab Dose 4 | Phase 1: Zalifrelimab Dose 5 | Phase 2: Zalifrelimab
All-Cause Mortality (participants affected / at risk) | 2/5 | 1/3 | 6/10 | 6/15 | 3/5 | 26/51
Serious Adverse Events (participants affected / at risk) | 2/5 | 2/3 | 5/10 | 9/15 | 3/5 | 23/51
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3 | 10/10 | 15/15 | 5/5 | 48/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Zalifrelimab Dose 1 (N=5) | Phase 1: Zalifrelimab Dose 2 (N=3) | Phase 1: Zalifrelimab Dose 3 (N=10) | Phase 1: Zalifrelimab Dose 4 (N=15) | Phase 1: Zalifrelimab Dose 5 (N=5) | Phase 2: Zalifrelimab (N=51)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1
Autoimmune colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oesophagael obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Blood creatine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Immune-mediated pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Thrombotic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Phase 1: Zalifrelimab Dose 1 (N=5) | Phase 1: Zalifrelimab Dose 2 (N=3) | Phase 1: Zalifrelimab Dose 3 (N=10) | Phase 1: Zalifrelimab Dose 4 (N=15) | Phase 1: Zalifrelimab Dose 5 (N=5) | Phase 2: Zalifrelimab (N=51)
Nausea (Gastrointestinal disorders) | 1 | 1 | 4 | 5 | 3 | 14
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 2 | 7 | 2 | 13
Constipation (Gastrointestinal disorders) | 1 | 1 | 4 | 5 | 3 | 11
Vomiting (Gastrointestinal disorders) | 3 | 2 | 4 | 6 | 1 | 9
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 1 | 3 | 1 | 8
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 1 | 5
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 3
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Autoimmune colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mesenteric panniculitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Salivary gland pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 5 | 9 | 4 | 17
Pyrexia (General disorders) | 1 | 1 | 2 | 5 | 0 | 5
Oedema peripheral (General disorders) | 0 | 0 | 1 | 3 | 1 | 8
Chills (General disorders) | 0 | 0 | 1 | 1 | 1 | 2
Chest pain (General disorders) | 2 | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 1 | 1
Malaise (General disorders) | 0 | 0 | 1 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
Oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Generalised oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mass (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 2 | 6 | 1 | 5
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 2 | 6 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 6 | 0 | 2
Weight decreased (Investigations) | 0 | 0 | 2 | 1 | 1 | 5
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 4 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 3 | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 2 | 0 | 2
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 2 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Lymph node palpable (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 2 | 5 | 0 | 11
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 5 | 0 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2 | 0 | 7
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 2 | 3 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 3 | 0 | 10
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 3 | 1 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 5 | 2 | 7
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 5 | 1 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0 | 6
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 5 | 0 | 8
Headache (Nervous system disorders) | 1 | 1 | 2 | 3 | 0 | 4
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 5 | 1 | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 2 | 1 | 0 | 3
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1
Abscess soft tissue (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urethral obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 4 | 1 | 2
Hypertension (Vascular disorders) | 0 | 1 | 2 | 0 | 1 | 3
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
Embolism (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 | 1 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 1 | 0 | 4
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 3
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 4
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 5
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 3
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/2 | 0/2 | 0/7 | 1/8 | 0/3 | 1/19 — Adverse event only affected female participants.
Pelvic discomfort (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/22/NCT02694822/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/22/NCT02694822/SAP_001.pdf